CLINICAL TRIAL: NCT04727710
Title: Testing the Effect of Mindfulness for Prostatectomy Outcomes (TEMPO)
Brief Title: Testing the Effect of Mindfulness for Prostatectomy Outcomes
Acronym: TEMPO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was held due to COVID19 and unable to enroll in virtual platform
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2018.129; HUM00152158 (Other: University of Michigan)
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Prostate Cancer
Keywords: Mindfulness
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 2: Couples-based mindfulness intervention (Experimental): Mindfulness-based intervention + Usual care
  Interventions: Behavioral: Mindfulness-based Intervention; Behavioral: Usual Care
- Part 2: Usual care (Active Comparator): Usual care
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — A self-directed, web-based mindfulness training. Investigators recommend one module a week for 6 weeks. Each module is approximately 1 hour long and consists of didactic components as well as meditation and mindfulness exercises.
  Arms: Part 2: Couples-based mindfulness intervention
Behavioral: Usual Care — Standard pre-operative survivorship seminar, offered monthly to all patients at Michigan Medicine about to undergo prostatectomy and their partners is aimed at promoting realistic expectations of prostatectomy outcomes, typical side effects, rehabilitation and emotional adjustment.

SUMMARY:
This research project has 2 parts: The first part of the research is to develop a couples-based group mindfulness intervention for men undergoing prostatectomy, with input from patients and their partners. The second part is the trial registered here, which will pilot the researchers' mindfulness intervention, developed in part 1, and observe any reduction of distress for men undergoing prostatectomy and their partners.

DETAILED DESCRIPTION:
In part 1 of this research, researchers developed a couples-based group mindfulness intervention for men undergoing prostatectomy, with input from patients and their partners. Three patients who had previously undergone prostatectomy, and had expressed interest in participating in future research endeavors, and their partners were recruited to inform the design of the intervention. This group of six stakeholders identified the types of distress experienced by newly diagnosed prostate cancer patients and their partners, as well as their favored intervention approaches. These stakeholders do participate in the intervention or control groups in part 2 of this study.

Researchers used thematic analysis to assess the type of distress identified by stakeholders as well as approaches favored by them. They mapped these themes on the available mindfulness approaches, identified in their review, to develop an intervention that best captures the concerns of prostate cancer survivors and partners.

Part 2 is the pilot study. Researchers will enroll 20 more couples (men who are planning to undergo radical prostatectomy and their partners) to participate in a pilot study of the intervention. The pilot study will have 2 cohorts (groups). Half of the couples will be randomly assigned to the mindfulness intervention (intervention group) and the other half will receive the usual care (control group). All participants in the intervention and control groups in part 2 of the study will be analyzed to determine the effects and feasibility of the intervention.

ELIGIBILITY:
Part 2--Pilot study:

Inclusion Criteria

* Patients aged 35 - 90 who are planning to undergo radical prostatectomy at University of Michigan Hospital
* Partners of these men, aged 18 and older

Exclusion Criteria:

* Participants cannot be less than 18 years of age

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change in level of distress assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form (SF) Anxiety | Change from baseline at 3 and 6 months post-prostatectomy
  This survey is administered as part of the patient's standard clinical care at University of Michigan. PROMIS SF Anxiety is an 8 item scale, each item is scored 1-5 where 1 is never and 5 is always. Higher scores indicate higher levels of anxiety.
Change in level of distress assessed using the PROMIS SF Depression. | Change from baseline at 3 and 6 months post-prostatectomy
  This survey is administered as part of the patient's standard clinical care at University of Michigan. PROMIS SF Depression is an 8 item scale, each item is scored 1-5 where 1 is never and 5 is always. Higher scores indicate higher levels of depression.
Change in level of distress assessed using the PROMIS SF Positive Affect and Well Being | Change from baseline at 3 and 6 months post-prostatectomy
  This survey is administered as part of the patient's standard clinical care at University of Michigan. PROMIS SF Positive Affect and Well Being is an 8 item scale, each item is scored 1-5 where 1 is never and 5 is always. Higher scores indicate higher levels of positive affect and well being.

SECONDARY OUTCOMES:
Change in salivary cortisol level (only patients will complete this, not partners) | Change from baseline at 3 months post-prostatectomy
  Saliva is collected through an at home collection kit that is mailed to the lab.
Change in level of distress assessed using the National Comprehensive Cancer Network (NCCN) Distress Thermometer | Change from baseline to 3 months post-prostatectomy
  The NCCN Distress Thermometer is a 1-item global screener of distress using a 0-10 scale with 10 being most distressed.
Change in level of distress assessed using the 5-facet Mindfulness Questionnaire (FFMQ) | Change from baseline at 3 months post-prostatectomy
  FFMQ is a 15 item self-reported assessment of mindfulness. Each item is scored 1-5, with higher scores indicating higher use of 5 key facets of mindfulness: Observing; Describing; Acting with awareness; Non-judging; Non-reactivity.
Change in urinary and sexual function assessed using Michigan Urological Surgery Improvement Collaborative (MUSIC) Expanded Prostate Cancer Index Composite (EPIC-26) | Change from baseline at 3 and 6 months post-prostatectomy
  MUSIC's EPIC-26 is a 26-item survey. Response options form a Likert scale, and multi-item scale scores are transformed linearly to a 0-100 scale, with higher scores representing higher levels of continence and better erectile function.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Herrel, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No